CLINICAL TRIAL: NCT05479448
Title: Predictive Factors for Treatment Response in Patients With Newly-diagnosed Polymyalgia Rheumatica and Giant Cell Arteritis
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Schweizerische Stiftung für die Erforschung der Muskelkrankheiten (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-00788; mu22Daikeler
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Polymyalgia Rheumatica (PMR); Giant Cell Arteritis (GCA)
Keywords: Large vessel vasculitis (LVV); Glucocorticoid receptor (GCR); glucocorticoid (GC); steroid-response; GCR expression levels; GCR sensitivity/responsiveness; prednisolone; prednisone; Swiss Clinical Quality Management in Rheumatic Diseases (SCQM); Glucocorticoid resistance; endogenous GC suppression
MeSH Terms: conditions — Polymyalgia Rheumatica; Giant Cell Arteritis; Glucocorticoid Receptor Deficiency | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection for cellular analyses (Immune subset composition, GCR expression, in vitro steroid responsiveness) — Biological material will be sampled at three time-points. The first time-point will be when patients have been treated with 15 mg of prednisone per day for at least 5 days. A second time-point will be after prednisone was successfully tapered and maintained at 5 mg per day for at least 5 days, a third time point will be 4 weeks after the stop of prednisone. Biosampling is done for cellular analyses, pharmacokinetics and hormone measurements.
Other: Data collection for exploratory analyses of endogenous steroid hormones — Concentrations of GC, MC, androgens and progestins will be determined and the suppression of cortisol and cortisone upon prednisone treatment will be analyzed.
Other: Data collection for correlation between clinical defined and lab defined GC responsivness — The time to first relapse, the cumulative steroid dose at 1 year after diagnosis, the need for treatment with steroid sparing agents and the GTI after 1 year will be correlated to the percentage of in vitro inhibition of cytokine concentration by dexamethasone treatment, to the prednisone/prednisolone ratio in plasma, to the percentage of endogenous GC suppression (plasma and urinary cortisol and cortisone) by prednisone treatment. Furthermore, correlations of steroid sensitivity with Mineralocorticoid (MC) and androgens will be investigated.
Other: Data collection for Prednisone metabolism — Plasma concentrations of prednisone and its active metabolite prednisolone will be quantified by liquid chromatography-tandem mass spectrometry (LC-MS/MS). If changes on prednisone/prednisolone are observed, the quantification of the 6-hydroxylated prednisone/prednisolone metabolites in 24 h urine samples will be performed to estimate their metabolism as well as the ratio of inactive to active GC.

SUMMARY:
This prospective study is to explore different predictive factors for response to steroid treatment in patients with PMR and/or GCA. It evaluates the association of endogenous GC suppression (plasma and urinary cortisol and cortisone) to the responsiveness of PMR/GCA to GCs.

DETAILED DESCRIPTION:
Polymyalgia rheumatica (PMR) and giant cell arteritis (GCA) are closely related inflammatory rheumatic diseases. The first-line treatment of both PMR and GCA are glucocorticoids (GC). In PMR, initial oral prednisone equivalent doses in between 10 and 25 mg/day are given. In contrast, GCA is usually treated with significantly higher steroid doses (starting dose 1 mg/kg body-weight) to prevent vascular complications.

The dose and duration of steroid treatment needed to control disease in patients with PMR and GCA vary and about half of the patients experience relapses, early upon GC dose tapering or after discontinuation of treatment. The reasons for the inter-individual differences in steroid-response are not known. Data from this controlled prospective study will help to identify subjects with GC resistance which would allow to use intensified treatment strategies (higher dose or alternative immune modulatory therapy) to overcome resistance. On the other hand, strong responsiveness to GC would provide a rational for rapid steroid tapering or treatment with lower doses, both resulting in reduced risk for GC related adverse events such as osteoporosis, infections, diabetes and mood disorders. Detailed understanding of the relation of individual GC signaling and GC metabolism with patients' response to steroid treatment will help to define steroid responder profiles. This prospective study is to explore different predictive factors for response to steroid treatment in patients with PMR and/or GCA.

At inclusion and at all follow-up visits, the clinical evaluation will be documented in the SCQM database. All participants with PMR will be treated according to our local treatment protocol: starting dose is 15 mg prednisone/d, tapered by 2.5 mg every second week once symptoms are controlled. After tapering to 10 mg/d, prednisone dose is further reduced by 2.5 mg every month.

All patients with GCA are treated according to published guidelines with prednisone starting at 1mg/kg body-weight followed by reduction to 0 mg at week 26 (GIACTA protocol).

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of PMR according to the 2012 provisional classification criteria and GCA according to published criteria
* Consent to participate in the SCQM database
* Treatment according to our standardized regimes

Exclusion Criteria:

* Treatment with Tocilizumab, MTX or other disease modifying medications at inclusion
* History of GCA and PMR in the past
* Inability to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting in the University Hospital Basel with newly diagnosed PMR according to the 2012 provisional classification criteria ) and patients with newly diagnosed GCA will be screened for inclusion. Final diagnosis of GCA is made either (i) if temporal artery biopsy is positive, (ii) if patients fulfill the 1989 ACR criteria, or (iii) if they fulfill at least 2/5 ACR criteria in combination with typical vasculitic ultrasound findings or vasculitic findings in other imaging methods.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Relapse (no/yes) of PMR/ GCA | Within one year after PMR/GCA diagnosis
  Relapse (no/yes) of PMR/ GCA (associated with endogenous cortisol levels under stable doses of 15 mg of prednisone). Relapse of GCA and or PMR is defined as intensification of immune-suppressive treatment due to symptoms, signs or laboratory values judged by the caring physician to be due to PMR or GCA.

SECONDARY OUTCOMES:
Cumulative steroid dose at 1 year after diagnosis | At 1 year after diagnosis
  Cumulative steroid dose at 1 year after diagnosis
Number of patients with Tocilizumab or other immunosuppressive/ biological treatment started within 1 year after diagnosis. | Within one year after PMR/GCA diagnosis
  Number of patients with Tocilizumab or other immunosuppressive/ biological treatment started within 1 year after diagnosis.
Number of patients with Methotrexate (MTX) treatment started within 1 year after diagnosis | Within one year after PMR/GCA diagnosis
  Number of patients with Methotrexate (MTX) treatment started within 1 year after diagnosis
Prednisone/prednisolone ratio in plasma | Within one year after PMR/GCA diagnosis
  Prednisone/prednisolone ratio in plasma
Glucocorticoid Toxicity Index (GTI) at 1 year after diagnosis | At 1 year after diagnosis
  Glucocorticoid Toxicity Index (GTI) at 1 year after diagnosis. The GTI is composed of 9 domains and measures the change in glucocorticoid toxicity between 2 points in time. The GTI can measure not only the worsening of glucocorticoid toxicity but also its improvement. The minimal clinically important difference for the GTI scores is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Daikeler, Prof. Dr. med., Principal Investigator — Department of Rheumatology University Hospital Basel
Locations (1):
- Department of Rheumatology University Hospital Basel, Basel, Switzerland